CLINICAL TRIAL: NCT03137069
Title: A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Controlled Pilot and Dose-Ranging Study of GDC-0853 in Patients With Refractory Chronic Spontaneous Urticaria (CSU).
Brief Title: A Study of GDC-0853 in Participants With Refractory Chronic Spontaneous Urticaria (CSU).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS39684; 2016-004624-35 (EudraCT Number)
Record Dates: First submitted 2017-04-28; First posted 2017-05-02 (Actual); Results first posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Urticaria
MeSH Terms: conditions — Urticaria | interventions — fenebrutinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1: Placebo (Placebo Comparator): Participants received matching placebo twice daily from Day 1 to 56.
  Interventions: Drug: Placebo
- Cohort 1: GDC-0853 200mg BID (Experimental): Participants received GDC-0853 200mg twice daily from Day 1 to 56.
  Interventions: Drug: GDC-0853
- Cohort 2: Placebo (Placebo Comparator): Participants received matching placebo up to twice daily from Day 1 to 56.
  Interventions: Drug: Placebo
- Cohort 2: GDC-0853 50mg QD (Experimental): Participants received GDC-0853 50mg once daily from Day 1 to 56.
  Interventions: Drug: GDC-0853
- Cohort 2: GDC-0853 150mg QD (Experimental): Participants received GDC-0853 150mg once daily from Day 1 to 56.
  Interventions: Drug: GDC-0853
- Cohort 2: GDC-0853 200mg BID (Experimental): Participants received GDC-0853 200mg twice daily from Day 1 to 56.
  Interventions: Drug: GDC-0853

INTERVENTIONS:
Drug: GDC-0853 — GDC-0853 will be administered orally at dosages of 50, 150 and 200mg to participants, as per the dosing schedules described above.
  Arms: Cohort 1: GDC-0853 200mg BID; Cohort 2: GDC-0853 150mg QD; Cohort 2: GDC-0853 200mg BID; Cohort 2: GDC-0853 50mg QD
Drug: Placebo — Matching Placebo will be administered orally, as per the dosing schedules described above.
  Arms: Cohort 1: Placebo; Cohort 2: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and pharmacokinetics of GDC-0853 compared with placebo in participants with Refractory Chronic Spontaneous Urticaria (CSU) already treated with anti-histamines. Participants have the option to enter the Open-Label Extension (OLE) study after completing the 8-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years, inclusive
* Diagnosis of chronic spontaneous urticaria (CSU) refractory to H1 antihistamines at the time of randomization
* Willing and able to complete an Urticaria Participant Daily eDiary for the duration of the study
* No evidence of active or latent or inadequately treated infection with tuberculosis (TB)
* Partcipants with a history of Bacille Calmette-Guérin (BCG) vaccination should be screened using the QuantiFERON-TB-Gold (QFT) test
* Only for participants currently receiving proton-pump inhibitors (PPIs) or H2 receptor antagonists (H2RAs): Treatment must be at a stable dose during the 2-week screening period prior to randomization and with a plan to remain at a stable dose for the duration of the study
* For women of childbearing potential: Agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least 4 weeks after the last dose of study drug. Women must refrain from donating eggs during this same period.

Exclusion Criteria:

* Treatment with omalizumab or other monoclonal antibody therapies used to treat CSU within 4 months prior to screening or primary nonresponse to omalizumab
* Use of a non-biologic investigational drug or participation in an investigational study with a non-biologic drug within 30 days prior to study drug administration on Day 1 (or within 5 half-lives of the investigational product, whichever is greater)
* Use of a biologic investigational therapy or participation in an investigational study involving biologic therapy within 90 days or 5 half-lives, whichever is greater, prior to study drug administration on Day 1
* Previous treatment with GDC-0853 or other Bruton's tyrosine kinase (BTK) inhibitors
* Participants whose urticaria is solely due to physical urticaria
* Other diseases with symptoms of urticaria or angioedema, including urticarial vasculitis, urticaria pigmentosa, erythema multiforme, mastocytosis, hereditary or acquired angioedema, lymphoma, or leukemia
* Atopic dermatitis, bullous pemphigoid, dermatitis herpetiformis, or other skin disease associated with itch such as psoriasis
* Routine doses of the following medications within 30 days prior to screening: systemic or cutaneous (topical) corticosteroids (prescription or over the counter), hydroxychloroquine, methotrexate, cyclosporine, or cyclophosphamide
* Prior utilization of intravenous (IV) steroids for treatment of laryngeal angioedema
* Intravenous immunoglobulin G (IV IG) or plasmapheresis within 30 days prior to screening
* History of anaphylactic shock without clearly identifiable avoidable antigen
* Hypersensitivity to GDC-0853 or any component of the formulation
* Major surgery within 8 weeks prior to screening or surgery planned prior to end of study (12 weeks after randomization)
* Require any prohibited concomitant medications
* History of live attenuated vaccine within 6 weeks prior to randomization or requirement to receive these vaccinations at any time during study drug treatment
* Evidence of clinically significant cardiac, neurologic, psychiatric, pulmonary, renal, hepatic, endocrine, metabolic, or gastrointestinal (GI) disease that, in the investigator's opinion, would compromise the safety of the participant, interfere with the interpretation of the study results or otherwise preclude participant participation
* Current treatment with astemizole, terfenadine, and/or ebastine
* Uncontrolled disease states, such as asthma, psoriasis, or inflammatory bowel disease, where flares are commonly treated with oral or parenteral corticosteroids

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (27):
- United States (13):
  - Clinical Research Center of Alabama, LLC, Birmingham, Alabama
  - Allergy & Asthma Immunology Associates, Scottsdale, Arizona
  - Kern Allergy Med Clinic, Inc., Bakersfield, California
  - Southern California Research Center, Mission Viejo, California
  - Allergy & Asthma Consultants, Redwood City, California
  - Integrated Research Group Inc, Riverside, California
  - Integrated Research of Inland, Upland, California
  - New Horizon Research Center, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Vital Prospects Clinical Research Institute PC - CRN, Tulsa, Oklahoma
  - Asthma, Nasal Disease, and Allergy Research Center of New England, East Providence, Rhode Island
  - Center for Clinical Studies, Cypress, Texas
  - Timber Lane Allergy and Asthma Research, LLC, Burlington, Vermont
- Canada (8):
  - University of British Columbia, Vancouver, British Columbia
  - Private Practice - Dr. Jason Ohayon, Hamilton, Ontario
  - Lynde Institute for Dermatology, Markham, Ontario
  - Cheema Research, Mississauga, Ontario
  - Yang Medicine, Ottawa, Ontario
  - Gordon Sussman Clinical Research, Toronto, Ontario
  - Private Practice - Dr. Isabelle Delorme, Drummondville, Quebec
  - Centre de Recherche Applique En Allergie de Quebec, Québec, Quebec
- Germany (6):
  - Licca Clinical Research Institute, Augsburg
  - Charite Mitte; Klinik fur Dermatologie, Berlin
  - Universitätsklinikum Carl Gustav Carus, Klinik und Poliklinik für Augenheilkunde, Dresden
  - Hautarztpraxis Mahlow, Mahlow
  - Universitätsmedizin Johannes Gutenberg Universität, Mainz
  - Klinik für Haut- und Geschlechtskrankheiten, Universitätsklinikum Münster, Münster

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 21 centers in 3 countries.
Pre-assignment Details: A total of 134 participants were enrolled at 21 centers.
Period: Overall Study
Arm/Group | Cohort 1: Placebo | Cohort 1: GDC-0853 200mg BID | Cohort 2: Placebo | Cohort 2: GDC-0853 50mg QD | Cohort 2: GDC-0853 150mg QD | Cohort 2: GDC-0853 200mg BID
Started | 13 | 28 | 23 | 23 | 24 | 23
Completed | 12 | 22 | 20 | 17 | 22 | 21
Not Completed | 1 | 6 | 3 | 6 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 2 | 2 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 3 | 1 | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 1 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Data Entry Error | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Placebo | Cohort 1: GDC-0853 200mg BID | Cohort 2: Placebo | Cohort 2: GDC-0853 50mg QD | Cohort 2: GDC-0853 150mg QD | Cohort 2: GDC-0853 200mg BID | Total
Number analyzed (Participants) | 13 | 28 | 23 | 23 | 24 | 23 | 134
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.6 (11.0) | 41.3 (15.9) | 40.2 (14.7) | 45.0 (13.1) | 43.3 (16.7) | 44.3 (13.0) | 42.8 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 22 | 17 | 18 | 20 | 16 | 104
  Male | 2 | 6 | 6 | 5 | 4 | 7 | 30
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 0 | 1 | 5 | 2 | 5 | 2 | 15
  Not Hispanic or Latino | 13 | 27 | 16 | 21 | 19 | 20 | 116
  Not Stated | 0 | 0 | 1 | 0 | 0 | 1 | 2
  Unknown | 0 | 0 | 1 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 0 | 3 | 4 | 3 | 1 | 4 | 15
  Black or African American | 1 | 1 | 1 | 1 | 0 | 2 | 6
  White | 10 | 24 | 18 | 19 | 23 | 16 | 110
  Multiple | 2 | 0 | 0 | 0 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Urticaria Activity Score Over 7 Days (UAS7) at Day 57
Description: The Urticaria Activity Score (UAS) is a composite, diary-recorded score with numeric severity intensity ratings (0=none to 3=intense/severe) for the number of wheals (hives) and the intensity of the pruritus (itch) over the past 12 hours (twice daily). The daily UAS is calculated as the average of the morning and evening scores. The UAS7 is the weekly sum of the daily UAS, which is the composite score of the intensity of pruritus and the number of wheals. The maximum UAS7 value is 42. A higher score indicates worse disease. A negative change score (Day 57 score minus Baseline score) indicates improvement.
Time Frame: Baseline and Day 57
Population: The Modified Intent-To-Treat (mITT) Population was defined as all participants who received at least one dose of study treatment grouped for analysis according to the treatment arm to which they were randomized. Data presented below is only for participants included in the actual analysis.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Cohort 1: Placebo | Cohort 1: GDC-0853 200mg BID | Cohort 2: Placebo | Cohort 2: GDC-0853 50mg QD | Cohort 2: GDC-0853 150mg QD | Cohort 2: GDC-0853 200mg BID
Number analyzed (Participants) | 12 | 22 | 20 | 19 | 22 | 21
Score on a Scale | -19.16 (13.49) | -24.05 (9.74) | -11.25 (10.81) | -15.69 (14.25) | -17.05 (10.19) | -21.80 (14.80)
Statistical Analysis 1: Comparison: Cohort 1: Placebo vs Cohort 1: GDC-0853 200mg BID; Test type: Superiority; p = 0.0559, Mixed Models Analysis; Covariates included were region, treatment group, visit, and visit by treatment group interaction; Least Squares Mean Difference = -7.02, 90% CI 2-sided [-13.01 to -1.03]
Statistical Analysis 2: Comparison: Cohort 2: Placebo vs Cohort 2: GDC-0853 50mg QD; Test type: Superiority; p = 0.8892, Mixed Models Analysis; Covariates included were region, treatment group, visit, and visit by treatment group interaction; Least Squares Mean Difference = -0.51, 90% CI 2-sided [-6.60 to 5.58]
Statistical Analysis 3: Comparison: Cohort 2: Placebo vs Cohort 2: GDC-0853 150mg QD; Test type: Superiority; p = 0.0717, Mixed Models Analysis; Covariates included were region, treatment group, visit, and visit by treatment group interaction; Least Squares Mean Difference = -6.43, 90% CI 2-sided [-12.29 to -0.57]
Statistical Analysis 4: Comparison: Cohort 2: Placebo vs Cohort 2: GDC-0853 200mg BID; Test type: Superiority; p = 0.0097, Mixed Models Analysis; Covariates included were region, treatment group, visit, and visit by treatment group interaction; Least Squares Mean Difference = -9.53, 90% CI 2-sided [-15.50 to -3.55]

2. Secondary Outcome: Percentage of Participants Who Are Well-Controlled (UAS7 ≤ 6)
Description: The Urticaria Activity Score (UAS) is a composite, diary-recorded score with numeric severity intensity ratings (0=none to 3=intense/severe) for the number of wheals (hives) and the intensity of the pruritus (itch) over the past 12 hours (twice daily). The daily UAS is calculated as the average of the morning and evening scores. The UAS7 is the weekly sum of the daily UAS, which is the composite score of the intensity of pruritus and the number of wheals. The maximum UAS7 value is 42. A higher score indicates worse disease. Participants with UAS7 score ≤6 are considered well controlled.
Time Frame: Day 57
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort 1: Placebo | Cohort 1: GDC-0853 200mg BID | Cohort 2: Placebo | Cohort 2: GDC-0853 50mg QD | Cohort 2: GDC-0853 150mg QD | Cohort 2: GDC-0853 200mg BID
Number analyzed (Participants) | 13 | 28 | 23 | 23 | 24 | 23
Percentage of Participants | 30.8 | 57.1 | 21.7 | 34.8 | 45.8 | 56.5
Statistical Analysis 1: Comparison: Cohort 1: Placebo vs Cohort 1: GDC-0853 200mg BID; Test type: Superiority; p = 0.1087, Cochran-Mantel-Haenszel; Stratified by region
Statistical Analysis 2: Comparison: Cohort 2: Placebo vs Cohort 2: GDC-0853 50mg QD; Test type: Superiority; p = 0.3418, Cochran-Mantel-Haenszel; Stratified by region
Statistical Analysis 3: Comparison: Cohort 2: Placebo vs Cohort 2: GDC-0853 150mg QD; Test type: Superiority; p = 0.0459, Cochran-Mantel-Haenszel; Stratified by region
Statistical Analysis 4: Comparison: Cohort 2: Placebo vs Cohort 2: GDC-0853 200mg BID; Test type: Superiority; p = 0.0190, Cochran-Mantel-Haenszel; Stratified by region

3. Secondary Outcome: Change From Baseline in the UAS7 at Day 29
Description: The Urticaria Activity Score (UAS) is a composite, diary-recorded score with numeric severity intensity ratings (0=none to 3=intense/severe) for the number of wheals (hives) and the intensity of the pruritus (itch) over the past 12 hours (twice daily). The daily UAS is calculated as the average of the morning and evening scores. The UAS7 is the weekly sum of the daily UAS, which is the composite score of the intensity of pruritus and the number of wheals. The maximum UAS7 value is 42. A higher score indicates worse disease. A negative change score (Day 29 score minus Baseline score) indicates improvement.
Time Frame: Baseline and Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Cohort 1: Placebo | Cohort 1: GDC-0853 200mg BID | Cohort 2: Placebo | Cohort 2: GDC-0853 50mg QD | Cohort 2: GDC-0853 150mg QD | Cohort 2: GDC-0853 200mg BID
Number analyzed (Participants) | 13 | 24 | 21 | 19 | 23 | 21
Score on a Scale | -9.69 (10.70) | -22.15 (10.33) | -9.05 (9.82) | -16.97 (14.31) | -13.75 (12.93) | -21.69 (16.22)
Statistical Analysis 1: Comparison: Cohort 1: Placebo vs Cohort 1: GDC-0853 200mg BID; Test type: Superiority; p = 0.0010, Mixed Models Analysis; Covariates included were region, treatment group, visit, and visit by treatment group interaction; Least Squares Mean Difference = -12.88, 90% CI 2-sided [-18.94 to -6.82]
Statistical Analysis 2: Comparison: Cohort 2: Placebo vs Cohort 2: GDC-0853 50mg QD; Test type: Superiority; p = 0.4565, Mixed Models Analysis; Covariates included were region, treatment group, visit, and visit by treatment group interaction; Least Squares Mean Difference = -2.83, 90% CI 2-sided [-9.11 to 3.46]
Statistical Analysis 3: Comparison: Cohort 2: Placebo vs Cohort 2: GDC-0853 150mg QD; Test type: Superiority; p = 0.1711, Mixed Models Analysis; Covariates included were region, treatment group, visit, and visit by treatment group interaction; Least Squares Mean Difference = -5.03, 90% CI 2-sided [-11.10 to 1.03]
Statistical Analysis 4: Comparison: Cohort 2: Placebo vs Cohort 2: GDC-0853 200mg BID; Test type: Superiority; p = 0.0050, Mixed Models Analysis; Covariates included were region, treatment group, visit, and visit by treatment group interaction; Least Squares Mean Difference = -10.76, 90% CI 2-sided [-16.97 to -4.56]

4. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An Adverse Event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An Adverse Event can therefore be any unfavorable and unintended sign (including abnormal laboratory values or abnormal clinical test results), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as Adverse Events.
Time Frame: Baseline up until 4 weeks after the last dose of study drug (up to 2 years, 5 months).
Population: The Safety-evaluable population was defined as all participants who received at least one dose of study drug with participants grouped according to their actual treatment. Due to a data entry error, one participant in the (Cohort 2: Placebo) arm was inadvertently analysed in the (Cohort 2: GDC-0853 200 mg BID) arm.
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort 1: Placebo | Cohort 1: GDC-0853 200mg BID | Cohort 2: Placebo | Cohort 2: GDC-0853 50mg QD | Cohort 2: GDC-0853 150mg QD | Cohort 2: GDC-0853 200mg BID
Number analyzed (Participants) | 13 | 28 | 22 | 23 | 24 | 24
Percentage of Participants | 61.5 | 71.4 | 54.5 | 60.9 | 66.7 | 58.3

5. Secondary Outcome: Plasma Concentrations of Fenebrutinib (GDC-0853) at Specified Timepoints
Description: Plasma Concentration Data for fenebrutinib (GDC-0853) will be tabulated and summarised by visits. Descriptive summary statistics for Arithmetic Mean and Standard Deviation will be presented. Please note that the Placebo Cohorts were not evaluated for this Outcome Measure.
Time Frame: Days 1, 8 and 57.
Population: The PK-evaluable population was defined as all participants who received at least one dose of fenebrutinib (GDC-0853) and had at least 1 evaluable post-dose PK sample. Participants who received incorrect therapy different from the intended therapy were summarized in the group according to the therapy actually received.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: GDC-0853 200mg BID | Cohort 2: GDC-0853 50mg QD | Cohort 2: GDC-0853 150mg QD | Cohort 2: GDC-0853 200mg BID
Number analyzed (Participants) | 28 | 23 | 24 | 23
ng/mL
  Day 1 | NA (NA) — No drug administered at this timepoint. | NA (NA) — No drug administered at this timepoint. | NA (NA) — No drug administered at this timepoint. | NA (NA) — No drug administered at this timepoint.
  Day 8 | 378 (389) | 38.5 (36.9) | 178 (237) | 424 (385)
  Day 57 | 283 (315) | 19.6 (26.3) | 24.7 (17.7) | 219 (293)

ADVERSE EVENTS:
Time Frame: Baseline up until 4 weeks after the last dose of study drug (up to 2 years, 5 months).
Description: One participant in Cohort 2 was randomized into the Placebo arm (Cohort 2: Placebo) and received the Placebo treatment in the study. However due to a data entry error, this participant was inadvertently analysed in the (Cohort 2: GDC-0853 200 mg BID) arm in the Safety-evaluable population.
Arm/Group | Cohort 1: Placebo | Cohort 1: GDC-0853 200mg BID | Cohort 2: Placebo | Cohort 2: GDC-0853 50mg QD | Cohort 2: GDC-0853 150mg QD | Cohort 2: GDC-0853 200mg BID
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/28 | 0/22 | 0/23 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/13 | 3/28 | 0/22 | 0/23 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 8/13 | 16/28 | 7/22 | 7/23 | 13/24 | 12/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Placebo (N=13) | Cohort 1: GDC-0853 200mg BID (N=28) | Cohort 2: Placebo (N=22) | Cohort 2: GDC-0853 50mg QD (N=23) | Cohort 2: GDC-0853 150mg QD (N=24) | Cohort 2: GDC-0853 200mg BID (N=24)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERIORBITAL CELLULITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEPATIC ENZYME INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Placebo (N=13) | Cohort 1: GDC-0853 200mg BID (N=28) | Cohort 2: Placebo (N=22) | Cohort 2: GDC-0853 50mg QD (N=23) | Cohort 2: GDC-0853 150mg QD (N=24) | Cohort 2: GDC-0853 200mg BID (N=24)
VISION BLURRED (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
CHILLS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
FEELING ABNORMAL (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EYE INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 3 (3) | 7 (9) | 1 (1) | 3 (3) | 3 (4) | 3 (4)
TOOTH INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
BONE CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
WEIGHT DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 3 (3) | 4 (5) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
CHRONIC SPONTANEOUS URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 1 (1) | 1 (2) | 2 (3) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) | 2 (2) | 3 (3) | 4 (4) | 5 (5)

LIMITATIONS AND CAVEATS:
Recruitment was stopped after an interim analysis of Cohort 2 based on pre-specified internal criteria.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-09): https://cdn.clinicaltrials.gov/large-docs/69/NCT03137069/Prot_SAP_000.pdf